CLINICAL TRIAL: NCT04805944
Title: Gut Microbiota, Pharmacogenetics and Integrase Strand Transfer Inhibitors Response
Brief Title: Gut Microbiota, PGx and INSTIs Response
Status: Completed | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: INSTI
Record Dates: First submitted 2021-03-08; First posted 2021-03-18 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: HIV Infections
Keywords: integrase strand transfer inhibitors; hiv; dolutegravir; bictegravir
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — dolutegravir; bictegravir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Stools
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- DTG treated (A): 80 HIV-infected adults treated with dolutegravir (as a component of their usual provider-prescribed antiretroviral regimen)
  Interventions: Drug: Dolutegravir
- BIC treated (B): 30 HIV-infected adults treated with bictegravir (as a component of their usual provider-prescribed antiretroviral regimen)
  Interventions: Drug: Bictegravir
- DTG discontinued due to neuropsychiatric adverse event (C): 50 HIV-infected adults having stopped dolutegravir due to neuropsychiatric adverse effects (insomnia, depression, anxiety)
  Interventions: Drug: Dolutegravir
- Shifting to DTG (D): 20 virally controlled and immunologically functional HIV-infected adults shifting (as per standard care) from another ARV class to an antiretroviral regimen containing dolutegravir
  Interventions: Drug: Dolutegravir
- Shifting to BIC (E): 20 virally controlled and immunologically functional HIV-infected adults shifting (as per standard care) from another ARV class to an antiretroviral regimen containing bictegravir
  Interventions: Drug: Bictegravir

INTERVENTIONS:
Drug: Dolutegravir — Dolutegravir treated patients will be included and samples (blood for pharmacokinetic, pharmacogenetic et metabolite profiling, stools for microbiota profiling) drawn at follow-up.
  Groups: DTG treated (A)
Drug: Bictegravir — Bictegravir treated patients will be included and samples (blood for pharmacokinetic, pharmacogenetic and metabolite profiling, stools for microbiota profiling) drawn at follow-up.
  Groups: BIC treated (B)
Drug: Dolutegravir — Patient having discontinued dolutegravir will be included and samples (blood for pharmacogenetic and metabolite profiling, stools for microbiota profiling) drawn at follow-up.
  Groups: DTG discontinued due to neuropsychiatric adverse event (C)
Drug: Dolutegravir — Patients starting dolutegravir will be included and sampled both before (blood for pharmacogenetic and metabolite profiling, stools for microbiota profiling) and after (blood for pharmacokinetic and metabolite profiling, stools for microbiota profiling) the start of dolutegravir
  Groups: Shifting to DTG (D)
Drug: Bictegravir — Patients starting bictegravir will be included and sampled both before (blood for pharmacogenetic and metabolite profiling, stools for microbiota profiling) and after (blood for pharmacokinetic and metabolite profiling, stools for microbiota profiling) the start of bictegravir
  Groups: Shifting to BIC (E)

SUMMARY:
This is an interventional phase IV trial enrolling HIV-infected patients treated by dolutegravir or bictegravir-based combined antiretroviral therapy, and patients with a planned shift to a dolutegravir or bictegravir-based combined antiretroviral therapy, that aims at understanding the individual response to dolutegravir and bictegravir, in terms of efficacy and toxicity.

DETAILED DESCRIPTION:
The main objective of our research project is to better define the inter-individual variability in terms of clinical and biological response towards Integrase Strand Transfer Inhibitors, an important ARV drug class used in the treatment of HIV infection. We aim at identifying predictors of drug efficacy and toxicity, which are eagerly awaited by clinicians as INSTIs are now prescribed worldwide and concerns about previously unidentified side effects are emerging.

The specific objectives of the project are:

* To study the impact of genetic polymorphisms in selected pharmacogenes (including genes coding for biotransformation enzymes and transport proteins) on INSTIs PK parameters and biomarkers relevant for TDM, such as trough (C0) and intracellular (IC) concentrations.
* To determine whether genetic polymorphisms in selected pharmacogenes might affect INSTIs efficacy, as assessed by the measurement of the viral load.
* To address the important question of the pathophysiological mechanisms lying behind the two main side effects of INSTIs, namely neuropsychiatric adverse events and abnormal weight gain.
* To describe how INSTIs affect the gut microbiome of treated patients, and to determine in turn how and by which pathways the gut microbiome might influence the clinical response (i.e. efficacy and toxicity) to INSTIs.

ELIGIBILITY:
Inclusion will be proposed to:

* HIV infected adult patient regularly followed at Centre de reference HIV of CUSL and currently treated by 50mg OD of DTG (n=80) or 50mg OD of BIC (n=30).
* Virally controlled immunologically functional HIV infected adult patient regularly followed at Centre de reference HIV of CUSL and shifting from another ARV class to a treatment containing 50mg OD of DTG (n=20) or 50mg OD of BIC (n=20).
* HIV infected adult patient retrospectively identified as having stopped standard dosage of DTG (ie. 50mg OD) due to NPAE (insomnia, depression, anxiety) (n=50). Identification will be based on the interrogation of our prospective clinical database.

Exclusion Criteria:

* Pregnancy at the time of inclusion or expected pregnancy within 12 months, for patients treated by DTG or BIC during the study
* Liver failure (Child-Pugh A, B or C)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited among regularly HIV-infected patients regularly followed at the Centre de Prise en charge VIH of Cliniques universitaires Saint-Luc - UCLouvain
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Dolutegravir and bictegravir through concentration | 24 hours post last dose
  Measurement of drug through concentration for groups A, B, D and E
Dolutegravir and bictegravir intracellular concentration | 24 hours post last dose
  Measurement of drug intracellular concentration for groups A, B, D and E
Viral replication | At least 3 months after the initiation of DTG/BIC
  Viral replication measured for groups A, B, D and E
Microbiota profile under treatment | At least 6 months after the initiation of DTG/BIC
  Determination microbiota profile for groups A, B, C, D and E
Change of microbiota profile | Baseline and at 6 months
  Change from baseline microbiota profile at 6 month after treatment initiation, for groups D and E
Change in weight | Through study completion, an average of 1 year
  Overall weight change between treatment initiation through study completion
Psychometric evaluation (Symptom-checklist-90-R) | At least 3 months after the initiation of DTG/BIC
  Psychometric evaluation through Symptom-checklist-90-R questionnaire, for groups A and B.
  The mean scores of each of the 10 subscales of Symptom-checklist-90-R will be calculated. A global severity index is computed as the average score of all 90 items. A higher score indicates a worse outcome.
Change of psychometric evaluation (Symptom-checklist-90-R) | Baseline and at 6 months
  Change from baseline Symptom-checklist-90-R at 6 month after treatment initiation, for groups D and E.
  The mean scores of each of the 10 subscales of Symptom-checklist-90-R will be calculated. A global severity index is computed as the average score of all 90 items. A higher score indicates a worse outcome.
Psychometric evaluation (Pittsburgh Sleep Quality Index) | At least 3 months after the initiation of DTG/BIC
  Psychometric evaluation through Pittsburgh Sleep Quality Index questionnaire, for groups A and B.
  Pittsburgh Sleep Quality Index scores answers from 0 to 21. A higher score means a worse outcome.
Change of psychometric evaluation (Pittsburgh Sleep Quality Index) | Baseline and at 6 months
  Change from baseline Pittsburgh Sleep Quality Index at 6 month after treatment initiation, for groups D and E.
  Pittsburgh Sleep Quality Index scores answers from 0 to 21. A higher score means a worse outcome.
Psychometric evaluation (Pichot's fatigue scale) | At least 3 months after the initiation of DTG/BIC
  Psychometric evaluation through Pichot's fatigue scale questionnaire, for groups A and B.
  Pichot's fatigue scale scores answers between 0 and 32. A higher score means a worse outcome.
Change of psychometric evaluation (Pichot's fatigue scale) | Baseline and at 6 months
  Change from baseline Pichot's fatigue scale at 6 month after treatment initiation, for groups D and E.
  Pichot's fatigue scale scores answers between 0 and 32. A higher score means a worse outcome.
Psychometric evaluation (Hospital Anxiety and Depression Scale) | At least 3 months after the initiation of DTG/BIC
  Psychometric evaluation through Hospital Anxiety and Depression Scale questionnaire, for groups A and B.
  Hospital Anxiety and Depression Scale scores answers between 0 and 21 for its two compoinents, anxiety and depression. A higher score means a worse outcome.
Change of psychometric evaluation (Hospital Anxiety and Depression Scale) | Baseline and at 6 months
  Change from baseline Hospital Anxiety and Depression Scale at 6 month after treatment initiation, for groups D and E.
  Hospital Anxiety and Depression Scale scores answers between 0 and 21 for its two compoinents, anxiety and depression. A higher score means a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Leïla Belkhir, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc; UCLouvain/IREC/LTAP
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

REFERENCES:
- [Derived] De Greef J, Nguyen KN, Van Hul M, Puel A, Yombi JC, Vandercam B, Vincent A, Elens L, Belkhir L, Haufroid V, Cani PD. Associations between weight gain, integrase inhibitors antiretroviral agents, and gut microbiome in people living with HIV: a cross-sectional study. Sci Rep. 2025 Jul 2;15(1):22603. doi: 10.1038/s41598-025-06500-0. PMID 40592975